CLINICAL TRIAL: NCT01153308
Title: Outcomes of Bariatric Surgery (UMMMC Bariatric Surgery Registry)
Brief Title: Outcomes of Bariatric Surgery/UMMMC Bariatric Surgery Registry
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: H-11612
Record Dates: First submitted 2010-03-21; First posted 2010-06-30 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Obesity; Weight Loss; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric Surgery Patients: Bariatric Surgery patients at UMass Memorial Medical Center
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — This is an Observational study

SUMMARY:
The purpose of this registry is to monitor and evaluate the efficacy, as well as safety, of bariatric surgery performed at UMass Memorial Medical Center, including laparoscopic gastric bypass surgery and laparoscopic gastric banding, in the surgical treatment of morbid obesity and associated co-morbidities such as type 2 diabetes, sleep apnea and cardiovascular disease.

DETAILED DESCRIPTION:
See brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for Bariatric Surgery @ UMMMC

Exclusion Criteria:

* Not scheduled for Bariatric Surgery @ UMMMC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UMMMC Bariatric Surgery Patients
Sampling Method: Non-Probability Sample
Enrollment: 4785 (Actual)
Dates: Start 2005-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Weight Loss after surgery | Preop, Postop, Six Months, and Annually
  Baseline weight is recorded preoperatively. Time points after surgery when weight is recorded are two weeks, six weeks, 6 months, 1 year, 18 months, 2 years, then annually on the anniversary date of surgery.

SECONDARY OUTCOMES:
Resolution of Co-morbidities, such as Type 2 Diabetes, Sleep Apnea, Hypertension | Preop, Postop, Six Months, Annually
  Preoperatively co-morbidities of morbid obesity are recorded as well as treatment (ie: medications, CPAP machine). Resolution of co-morbidities postoperatively is measured/recorded for example by blood tests, sleep study, as well as changes or discontinuation of medications &/or interventions.

CONTACTS AND LOCATIONS:
Overall Officials: John J Kelly, MD, Principal Investigator — University of Massachusetts Medical School and UMass Memorial Medical Center
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- See also: UMass Memorial Medical Center — http://www.umassmemorial.org